CLINICAL TRIAL: NCT03256747
Title: Effects of Neuromuscular Electrical Stimulation on Glucose Levels and Glucose Variability in Patients With Type 2 Diabetes: a Randomized Clinical Trial
Brief Title: Effects of Neuromuscular Electrical Stimulation on Glucose Variability in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68437417.0.0000.5327
Record Dates: First submitted 2017-08-07; First posted 2017-08-22 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: GCMS record will be coded and analyzed by a blinded investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES group (Experimental): NMES will be placed at the knee extensors, with maximal intensity tolerance evaluated by to induce visible contractions.
  Interventions: Device: NMES
- NMES-placebo group (Placebo Comparator): NMES-placebo will be placed at the knee extensors, with minimal intensity to provide a sensory stimulus, but insufficient to elicit a tetanic muscular contraction.
  Interventions: Device: NMES-placebo

INTERVENTIONS:
Device: NMES — NMES will be placed at the knee extensors. Stimulation frequency will be 20 Hz. Pulse width will be 0.5 milliseconds and the contraction time will be 10 seconds (TON: 10s) with a 5-second rest interval (TOFF: 5s). Total time application will be 60 minutes. Intensity will be adjusted individually, taking into account the patient's ability to promote the full knee extension and comfort during contractions.
  Arms: NMES group
Device: NMES-placebo — NMES-placebo will be placed at the knee extensors. Stimulation frequency will be 20 Hz. Pulse width will be 0.5 milliseconds and the contraction time will be 10 seconds (TON: 10s) with a 5-second rest interval (TOFF: 5s). Total time of application will be 60 minutes. Intensity will be adjusted with minimal intensity, utilized to provide a sensory stimulus, but insufficient to elicit a tetanic muscular contraction.
  Arms: NMES-placebo group

SUMMARY:
In patients with type 2 diabetes mellitus (T2DM) chronic hyperglycemia is the main cause of complications, promoting several micro and macrovascular damages. In order to understand other mechanisms that could have an impact on the development of these diabetic complications, the assessment of glycemic variability have been widely used. Glucose control can be achieved with multiple interventions, including exercise training. Some individuals, however, especially those with autonomic neuropathy, can have exercise intolerance. In this context, physical therapy proposes neuromuscular electrical stimulation (NMES) as a therapeutic that has been applied in research and clinical practice as an alternative to the training of patients who cannot perform conventional exercise. In patients with T2DM, NMES was shown to improve glycemic control and insulin sensitivity, but quality of these trials is poor. In addition, the effects of NMES on glycemic variability of T2DM patients have not yet been reported. The aim of this study is to evaluate the effects of NMES on glucose levels and glucose variability in patients with T2DM.

DETAILED DESCRIPTION:
Patients with T2DM will be recruited from outpatient clinic of the Hospital de Clinicas de Porto Alegre. Patients will be randomized to NMES session, with maximal intensity tolerance by to induce visible contractions or to NMES-placebo, with minimal intensity to provide a sensory stimulus, but insufficient to elicit a tetanic muscular contraction. Subjects will attend to research facility four times. On the first visit clinical, physical examination and autonomic evaluation (Ewing test) will be performed and a blood sample will be collected. On the second visit CGMS will be placed for glycemic variability evaluation. On the third visit NMES or NMES-placebo will be performed in a randomized way. On the fourth visit the CGMS will be removed. Blood pressure and heart rate will be evaluated during the protocol each 5 minutes and oxygenation tissue will be evaluated before, during and immediately after the protocol, through NIRS.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* HbA1c from 7,5 to 10%;
* Fasting plasma glucose lower to 250 mg/dL
* Drug therapy maintained for at least one month before inclusion in the study.

Exclusion Criteria:

* Insulin use;
* Pregnancy;
* Documented arrhythmia;
* Unstable angina;
* Chronic renal failure (GFR lower than 15 ml/min);
* Varicose vein problems;
* Clinical musculoskeletal disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Glucose levels | 48 hours
  Glucose levels will be assessed through continuous glucose monitoring (CGMS)

SECONDARY OUTCOMES:
Glucose variability | 48 hours
  Glucose variability will be assessed by CGMS 24 hours before, during the protocol and 24 hours after protocol.
Blood pressure | Each 5 minutes during intervention which will last 60 minutes.
  Will be evaluated through non-invasive oscillometric device.
Heart Rate | Each 5 minutes during intervention which will last 60 minutes.
  Will be evaluated through non-invasive oscillometric device.
Oxygenation tissue | Before, during and immediately after the intervention which will last 60 minutes.
  Will be evaluated through near infrared spectroscopy (NIRS).

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D Schaan, PhD, Principal Investigator — HCPA
Locations (1):
- Aline C P Macedo, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Brownlee M. The pathobiology of diabetic complications: a unifying mechanism. Diabetes. 2005 Jun;54(6):1615-25. doi: 10.2337/diabetes.54.6.1615. No abstract available. PMID 15919781
- [Background] Monnier L, Wojtusciszyn A, Colette C, Owens D. The contribution of glucose variability to asymptomatic hypoglycemia in persons with type 2 diabetes. Diabetes Technol Ther. 2011 Aug;13(8):813-8. doi: 10.1089/dia.2011.0049. Epub 2011 May 11. PMID 21561372
- [Background] Standards of Medical Care in Diabetes-2017: Summary of Revisions. Diabetes Care. 2017 Jan;40(Suppl 1):S4-S5. doi: 10.2337/dc17-S003. No abstract available. PMID 27979887
- [Background] Green S, Egana M, Baldi JC, Lamberts R, Regensteiner JG. Cardiovascular control during exercise in type 2 diabetes mellitus. J Diabetes Res. 2015;2015:654204. doi: 10.1155/2015/654204. Epub 2015 Mar 30. PMID 25918732
- [Background] Sbruzzi G, Ribeiro RA, Schaan BD, Signori LU, Silva AM, Irigoyen MC, Plentz RD. Functional electrical stimulation in the treatment of patients with chronic heart failure: a meta-analysis of randomized controlled trials. Eur J Cardiovasc Prev Rehabil. 2010 Jun;17(3):254-60. doi: 10.1097/HJR.0b013e328339b5a2. PMID 20560163
- [Background] Crowe L, Caulfield B. Aerobic neuromuscular electrical stimulation--an emerging technology to improve haemoglobin A1c in type 2 diabetes mellitus: results of a pilot study. BMJ Open. 2012 Jun 14;2(3):e000219. doi: 10.1136/bmjopen-2011-000219. Print 2012. PMID 22700835
- [Background] Joubert M, Metayer L, Prevost G, Morera J, Rod A, Cailleux A, Parienti JJ, Reznik Y. Neuromuscular electrostimulation and insulin sensitivity in patients with type 2 diabetes: the ELECTRODIAB pilot study. Acta Diabetol. 2015 Apr;52(2):285-91. doi: 10.1007/s00592-014-0636-5. Epub 2014 Aug 9. PMID 25107502